CLINICAL TRIAL: NCT03582774
Title: Phase III Randomized Multicenter Trial of 68Ga-PSMA-11 PET/CT Molecular Imaging for Prostate Cancer Salvage Radiotherapy Planning [PSMA-SRT]
Brief Title: Multicenter Randomized Trial of 68Ga-PSMA-11 PET/CT Based SRT After Radical Prostatectomy
Acronym: PSMA SRT
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Jonsson Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 18-000484; NCI-2018-01518 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); NUC MED 18-000484; 18-000484 (Other: UCLA / Jonsson Comprehensive Cancer Center); P30CA016042 (NIH)
Record Dates: First submitted 2018-06-19; First posted 2018-07-11 (Actual); Last update posted 2025-05-13 (Actual); Status verified 2025-05

CONDITIONS: Recurrent Prostate Carcinoma
Keywords: PSMA; PET/CT; salvage radiation therapy; randomized trial
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Practice Guidelines as Topic; Standard of Care; gallium 68 PSMA-11; 68Ga-DKFZ-PSMA-11; Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Arm I (standard of care) (Active Comparator): Participants receive standard of care SRT.
  Interventions: Other: Best Practice
- Arm II (68Ga-PSMA-11 PET/CT) (Experimental): Participants receive 68Ga-PSMA-11 IV and 50-100 minutes later undergo whole-body (skull base to mid-thighs) PET/CT. Participants then undergo SRT per the discretion of the treating radiation oncologist.
  Interventions: Procedure: Computed Tomography; Radiation: Gallium Ga 68-labeled PSMA-11; Procedure: Positron Emission Tomography

INTERVENTIONS:
Other: Best Practice — Undergo standard of care
  Other Names: standard of care; standard therapy
  Arms: Arm I (standard of care)
Procedure: Computed Tomography — Undergo PET/CT
  Other Names: CAT; CAT Scan; Computerized Axial Tomography; Computerized Tomography; CT; CT Scan; tomography
  Arms: Arm II (68Ga-PSMA-11 PET/CT)
Radiation: Gallium Ga 68-labeled PSMA-11 — Given IV
  Other Names: (68)Ga labeled Glu-NH-CO-NH-Lys(Ahx)-HBED-CC; (68)Ga-labeled Glu-urea-Lys(Ahx)-HBED-CC; (68)Ga-PSMA Ligand Glu-urea-Lys(Ahx)-HBED-CC; (68)Gallium-PSMA Ligand Glu-urea-Lys(Ahx)-HBED-CC; (68Ga)Glu-urea-Lys(Ahx)-HBED-CC; 68Ga-DKFZ-PSMA-11; 68Ga-HBED-CC-PSMA; 68Ga-labeled Glu-NH-CO-NH-Lys(Ahx)-HBED-CC; 68Ga-PSMA; 68Ga-PSMA-11; 68Ga-PSMA-HBED-CC; [68Ga] Prostate-specific Membrane Antigen 11; [68Ga]GaPSMA-11; Ga PSMA; Ga-68 labeled DKFZ-PSMA-11; Ga-68 labeled PSMA-11; Gallium Ga 68 PSMA-11; Gallium-68 PSMA; Gallium-68 PSMA Ligand Glu-urea-Lys(Ahx)-HBED-CC; GaPSMA; PSMA-HBED-CC GA-68
  Arms: Arm II (68Ga-PSMA-11 PET/CT)
Procedure: Positron Emission Tomography — Undergo PET/CT
  Other Names: Medical Imaging, Positron Emission Tomography; PET; PET Scan; Positron Emission Tomography Scan; Positron-Emission Tomography; proton magnetic resonance spectroscopic imaging
  Arms: Arm II (68Ga-PSMA-11 PET/CT)

SUMMARY:
This phase III trial studies how well Gallium Ga 68-labeled PSMA-11 (68Ga-PSMA-11) positron emission tomography (PET)/computed tomography (CT) works in diagnosing participants with prostate cancer that has come back after surgery. 68Ga-PSMA-11 are taken up by cancer cells. Diagnostic procedures, such as PET/CT scans, may help find and diagnose prostate cancer and find out how far the disease has spread. Giving 68Ga-PSMA-11 with PET/CT may help doctors plan better for salvage radiation therapy in participants with recurrent prostate cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. Success rate of salvage radiation therapy (SRT) measured as biochemical progression-free survival after initiation of SRT.

SECONDARY OBJECTIVES:

I. Sub-group analysis of the primary endpoint (success rate of SRT) within the subgroup with baseline PSA ≥ 0.5 ng/ml II. 5-year biochemical progression-free survival rate (from date of randomization).

III. Metastasis free survival. IV. Initiation of additional salvage therapy after completion of SRT. V. Change in initial treatment intent.

OUTLINE: Participants are randomized to 1 of 2 arms.

ARM I: Participants receive standard of care SRT.

ARM II: Participants receive 68Ga-PSMA-11 intravenously (IV) and 50-100 minutes later undergo whole-body (skull base to mid-thighs) PET/CT. Participants then undergo SRT per the discretion of the treating radiation oncologist.

After conclusion of PET/CT, participants are followed up periodically for up to 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Histopathology proven prostate cancer.
* Planned SRT for recurrence after primary prostatectomy.
* Prostate-specific antigen (PSA) >= 0.1 ng/ml at time of enrollment.
* Willingness to undergo radiotherapy.
* Treating radiation oncologist intends to incorporate 68Ga-PSMA-11 PET/CT findings into the radiotherapy plan if patient undergoes 68Ga-PSMA-11 PET/CT.

Exclusion Criteria:

* Extra-pelvic metastasis on any imaging or biopsy.
* Androgen deprivation therapy (ADT) within 3 months before 68Ga-PSMA-11 PET/CT.
* Contraindications to radiotherapy (including active inflammatory bowel disease).
* Concurrent systemic therapy for prostate cancer with investigational agents.

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 193 (Estimated)
Dates: Start 2018-07-12 (Actual); Primary Completion 2026-07-12 (Estimated); Study Completion 2027-07-12 (Estimated)

PRIMARY OUTCOMES:
Success rate of salvage radiation therapy (SRT) | From date of initiation of SRT assessed up to 5 years
  Will be measured as biochemical progression-free survival after initiation of SRT. Will use a log rank test to compare progression free survival time between the two randomized treatment arms.

SECONDARY OUTCOMES:
Biochemical progression-free survival rate | From date of randomization assessed up to 5 years
  Will utilize Cox-proportional hazards regression models. These models will include terms for treatment as well as appropriate clinical/demographic covariates (e.g., androgen deprivation therapy [ADT], pelvic lymph node radiation therapy [LN RT], prostate specific antigen [PSA] doubling time, Gleason grade, T stage, age, etc). Residual analyses will be performed to evaluate the proportional hazards assumptions of the Cox model. As a sensitivity analysis, we will also consider survival models that can account for competing risks (ex. death from other causes).
Metastasis free survival | Up to 5 years
  Will utilize Cox-proportional hazards regression models. These models will include terms for treatment as well as appropriate clinical/demographic covariates (e.g., ADT, pelvic LN RT, PSA doubling time, Gleason grade, T stage, age, etc). Residual analyses will be performed to evaluate the proportional hazards assumptions of the Cox model. As a sensitivity analysis, we will also consider survival models that can account for competing risks (ex. death from other causes).
Initiation of additional salvage therapy after completion of SRT | Up to 5 years
  Will utilize Cox-proportional hazards regression models. These models will include terms for treatment as well as appropriate clinical/demographic covariates (e.g., ADT, pelvic LN RT, PSA doubling time, Gleason grade, T stage, age, etc). Residual analyses will be performed to evaluate the proportional hazards assumptions of the Cox model. As a sensitivity analysis, we will also consider survival models that can account for competing risks (ex. death from other causes).
Change in initial treatment intent | Up to 5 years
  Will utilize Cox-proportional hazards regression models. These models will include terms for treatment as well as appropriate clinical/demographic covariates (e.g., ADT, pelvic LN RT, PSA doubling time, Gleason grade, T stage, age, etc). Residual analyses will be performed to evaluate the proportional hazards assumptions of the Cox model. As a sensitivity analysis, we will also consider survival models that can account for competing risks (ex. death from other causes).

CONTACTS AND LOCATIONS:
Overall Officials: Jeremie Calais, Principal Investigator — UCLA / Jonsson Comprehensive Cancer Center
Locations (2):
- United States (2):
  - UCLA / Jonsson Comprehensive Cancer Center, Los Angeles, California
  - UCSF Medical Center-Mount Zion, San Francisco, California

REFERENCES:
- [Derived] Calais J, Armstrong WR, Kishan AU, Booker KM, Hope TA, Fendler WP, Elashoff D, Nickols NG, Czernin J. Update from PSMA-SRT Trial NCT03582774: A Randomized Phase 3 Imaging Trial of Prostate-specific Membrane Antigen Positron Emission Tomography for Salvage Radiation Therapy for Prostate Cancer Recurrence Powered for Clinical Outcome. Eur Urol Focus. 2021 Mar;7(2):238-240. doi: 10.1016/j.euf.2020.12.009. Epub 2020 Dec 30. PMID 33386288
- [Derived] Calais J, Czernin J, Fendler WP, Elashoff D, Nickols NG. Randomized prospective phase III trial of 68Ga-PSMA-11 PET/CT molecular imaging for prostate cancer salvage radiotherapy planning [PSMA-SRT]. BMC Cancer. 2019 Jan 7;19(1):18. doi: 10.1186/s12885-018-5200-1. PMID 30616601